CLINICAL TRIAL: NCT02026115
Title: Computerized PAINRelieveIt Protocol for Cancer Pain Control in Hospice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); JourneyCare Home Health & Hospice (Unknown); Rainbow Hospice (Other)
Responsible Party: Principal Investigator, Diana J. Wilkie, Adjunct Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2013-0986; IH-1304-6553 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2013-12-28; First posted 2014-01-01 (Estimated); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Pain
Keywords: cancer; hospice; pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual hospice care (Active Comparator): The usual care group will receive the typical hospice care and interact with PAINReportIt to provide data necessary for the analysis of study aims. They will use the tablet computer at baseline and at the study end and daily between. They also will have access to what looks like PAINUCope, but is really computer games so that they have similar attention with the computer as the experimental group. For ethical purposes, we will provide a PAINReportIt Summary to their hospice nurses to have access to their pain assessment information, something we did not do in previous studies focused on efficacy of the interventions.
  Interventions: Behavioral: PAINReportIt
- PAINRelieveIt (experimental group) (Experimental): We will use Nursing Consult LLC's PAINRelieveIt software that includes: (1) PAINReportIt that has screens to collect pain, medications, and misconception data; (2) the intervention for the nurse clinicians, PAINConsultN; and (3) the intervention for the patients and lay caregiver, PAINUCope. This innovative, new program is the first computerized, multi-dimensional, self-report measure of pain with clinician decision support for analgesic prescriptions and multimedia patient education tailored to the patient's misconceptions and pain. Prototype versions of PAINConsultN and PAINUCope were tested in recently completed studies among outpatients with cancer and patients with sickle cell disease in outpatient, emergency and hospital settings.
  Interventions: Behavioral: PAINReportIt; Behavioral: PAINConsultN; Behavioral: PAINUCope

INTERVENTIONS:
Behavioral: PAINReportIt — PAINReportIt is a software program developed with an electronic McGill Pain Questionnaire (MPQ) and now includes questions about analgesics used by patients and a shortened version of the pain Barriers Questionnaire (BQ). It is designed as an interactive, touch screen way to assess pain. It can be self-administered and requires little or no patient computer experience and little or no provider time. The patient can read instructions on-screen and practice all types of selection responses found the program. Directions from the paper tools were modified to address the touch screen method of recording responses. The copyright is owned by Dr. Ronald Melzack for the MPQ and Dr. Sandra Ward for the BQ. Both individuals authorized the modifications, format, and computerized use of the tools.
  Other Names: PAINRelieveIt's PAINReportIt
Behavioral: PAINConsultN — PAINConsultN for hospice nurses. Our previous studies support the feasibility and clinical effect of PAINConsultN. This narrative and graphic tool provides decision support for the nurse's clinical decisions regarding management of the patient's pain. Based on the PAINReportIt output and published cancer pain guidelines, PAINConsultN generates an algorithm-based consultation report with a list of recommendations that could be useful to provide improved pain relief. If the patient's PAINReportIt output indicates the pain level is consistent with the patient's goals for pain management and represents no pain or a mild pain level, the consultation report acknowledges the therapy plan and reinforces its consistency with pain guidelines.
  Other Names: PAINRelieveIt's PANConsultN
  Arms: PAINRelieveIt (experimental group)
Behavioral: PAINUCope — We tested the PAINUCope piece of the intervention in 3 completed studies. PAINUCope is a multimedia, computer generated tool that gives tailored information to overcome patients' misconceptions about pain and help them engage in activities that help reduce their pain. PAINUCope focuses on 2 crucial aspects of pain management: 1) reporting cancer pain and 2) safe and effective use of pain medicines. The educational materials are written at a 6th grade reading level and presented as 21st Century best-practices, evidence-based facts or scripts for the person with cancer or sickle cell disease (in one study). The facts or scripts are customized to the patient's need for this type of health information. The patient's responses on PAINReportIt guide the specific information shared via PAINUCope.
  Other Names: PAINRelieveIt's PAINUCope
  Arms: PAINRelieveIt (experimental group)

SUMMARY:
The study purpose is to compare usual hospice care and PAINRelieveIt groups for effects on: (1) patient outcomes (analgesic adherence; worst pain intensity, satisfaction, and misconceptions) and lay caregiver outcome (pain misconceptions) in a diverse sample of 250 cancer patient-caregiver dyads receiving hospice care; and (2) nurse outcomes (obtained appropriate analgesics for patient) in a sample of hospice nurses. The investigators hypothesize that at posttest, controlling for pretest data and compared to the usual care group, the PAINRelieveIt group will: a) report decreased scores for worst pain intensity and pain misconceptions; b) have increased analgesic adherence (primary outcome); and c) have a larger proportion who report satisfaction with pain intensity and whose nurses obtained appropriate analgesics for the patients' pain.

DETAILED DESCRIPTION:
Unrelieved cancer pain at the end of life is a major health problem and is inconsistent with patient-centered goals for their last days. Building on a successful approach researched in outpatient oncology settings, the investigators propose a study testing PAINRelieveIt, a system-level intervention of computerized tools with patient-reported pain outcomes (in English, Spanish, Chinese languages), decision support for clinicians (English) and multimedia education tailored to each cancer patient and lay caregiver.

Using a 1-week pre-test/post-test randomized design in patients receiving home level hospice care provided by two Chicago-area hospices, we will compare effects of usual hospice care with PAINReportIt Summary and usual hospice care with PAINRelieveIt on pain outcomes. The tablet-based PAINRelieveIt includes valid and reliable pain tools (PAINReportIt), a summary of the patient's pain data with decision support for hospice nurses to obtain recommendations for algorithm-based analgesic therapies (PAINConsultN), and multimedia education tailored to the patient's and lay caregiver's pain management misconceptions (PainUCope). Patient's/caregiver's answers are automatically stored in an electronic database, from which the system generates a PAINReportIt Summary (usual hospice care control group); PAINConsultN and PainUCope (experimental group). All patients will receive usual hospice care. All patients/caregivers will complete PAINReportIt at pretest and 1-week later (posttest); patients also complete parts of PAINReportIt daily. Via daily e-mail updates, the control-group hospice nurses will receive a PAINReportIt Summary and experimental-group hospice nurses will receive a PAINConsultN. Additionally, experimental group patients/caregivers will view multimedia educational materials via PAINUCope to help patients report pain and adhere to prescribed analgesics.

Specific aims are to compare usual hospice care and PAINRelieveIt groups for effects on:

1. Patient outcomes (analgesic adherence; worst pain intensity, satisfaction, and misconceptions) and lay caregiver outcome (pain misconceptions) in a diverse sample of 250 cancer patient-caregiver dyads receiving hospice care.
2. Nurse outcomes (obtained appropriate analgesics for patient) in a sample of hospice nurses.

The investigators hypothesize that at posttest, controlling for pretest data and compared to the usual care group, the PAINRelieveIt group will: a) report decreased scores for worst pain intensity and pain misconceptions; b) have increased analgesic adherence (primary outcome); and c) have a larger proportion who report satisfaction with pain intensity and whose nurses obtained appropriate analgesics for the patients' pain.

Findings will guide future system-level research to implement PAINRelieveIt in a multi-site, longitudinal trial that will test the effect of disseminating this technology on clinical decisions for managing pain and patient/caregiver pain outcomes in a national sample of hospices. This approach offers improved pain control for dying patients and other populations.

ELIGIBILITY:
Inclusion Criteria:

Study inclusion criteria require that the patient: (1) be admitted to home care level of hospice service; (2) has a diagnosis of cancer; (3) has experienced worst pain in the past 24 hours >3 on a 0-10 scale; (4) speaks, reads and writes English, Spanish, or Chinese; (5) is > 18 years of age; 6) has a lay caregiver who is > 18 years of age and willing to participate; and (7) has a life expectancy of about 19 days at the time of study enrollment, as suggested by a Palliative Performance Scale (PPS)41 score of > 40.

The lay caregiver inclusion criteria require that the individual: (1) be designated as the primary lay caregiver for the participating patient during the 7-day study period; (2) speaks, reads and writes English, Spanish, or Chinese; and (3) is > 18 years of age.

The hospice nurse inclusion criteria require that the individual: (1) be assigned as the primary hospice nurse for the participating patient during the 7-day study period; (2) speaks, reads and writes English (since the PAINConsultN is in English) but may speak Spanish or Chinese for clinical care purposes; and (3) is > 18 years of age.

Exclusion Criteria:

* Patients and lay caregivers will be excluded if they: (1) are legally blind or deaf; or (2) have cognitive or physical impairments making it impossible to communicate or to complete study instruments at enrollment or any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana J Wilkie, PhD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Started | 170 | 92
Completed | 154 | 80
Not Completed | 16 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group) | Total
Number analyzed (Participants) | 154 | 80 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (14.4) | 69.5 (13.1) | 68.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 38 | 119
  Male | 73 | 42 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 14 | 42
  Not Hispanic or Latino | 126 | 66 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 25 | 81
  White | 71 | 44 | 115
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 22 | 11 | 33
Adherence Rate for Scheduled Opioids [Mean (Standard Deviation); unit: proportion of adherence (0-1)] — Analgesic adherence is derived from data regarding analgesics documented as prescribed (available to the patient as indicated from the medication list in the home) and analgesics consumed (from PAINReportIt). We calculate an analgesic adherence rate (dose reported as consumed divided by dose documented as prescribed) for all World Health Organization (WHO) analgesics (adjuvants, NSAIDs and non-opioids, and ATC and PRN Step 2 and Step 3 opioids).
  proportion of adherence (0-1) | 0.59 (0.33) | 0.66 (0.31) | 0.61 (0.33)
Worst Pain Intensity [Mean (Standard Deviation); unit: units on a scale (0-10)] — worst pain intensity in previous 24 hours measured on 0 to 10 scale where 0 means no pain and 10 means pain as bad as it can be.
  units on a scale (0-10) | 7.09 (2.29) | 6.99 (2.52) | 7.06 (2.37)
Least Pain Intensity [Mean (Standard Deviation); unit: units on a scale (0-10)] — least pain intensity in previous 24 hours measured on 0 to 10 scale where 0 means no pain and 10 means pain as bad as it can be.
  units on a scale (0-10) | 3.17 (2.40) | 3.09 (2.27) | 3.15 (2.35)
Current Pain Intensity [Mean (Standard Deviation); unit: units on a scale (0-10)] | 4.76 (2.72) | 4.64 (2.51) | 4.72 (2.64)
Satisfaction with Pain Level [Count of Participants; unit: Participants]
  Satisfied | 56 | 31 | 87
  Not sure | 16 | 10 | 26
  Not satisfied | 82 | 39 | 121
Pain Barrier -- Patient [Mean (Standard Deviation); unit: units on a scale (0-5)] — Misconceptions are measured with a computer version of the Barriers Questionnaire (BQ) with response options from 0 to 5 indicating the amount of agreement with statements about barriers to pain assessment or management. Items relate to communicating with the physician about pain, side effects of analgesics, concerns about addiction, tolerance, disease progression, and being perceived as a good patient. To improve the acceptability of the tool to patients with cancer, we reduced the tool to 13 items with demonstrated validity and reliability.
  units on a scale (0-5) | 2.75 (0.81) | 2.44 (0.86) | 2.64 (0.84)
Pain Barrier -- Caregiver [Mean (Standard Deviation); unit: units on a scale (0-5)] — Misconceptions are measured with a computer version of the Barriers Questionnaire (BQ) with response options from 0 to 5 indicating the amount of agreement with statements about barriers to pain assessment or management. Items relate to communicating with the physician about pain, side effects of analgesics, concerns about addiction, tolerance, disease progression, and being perceived as a good patient. To improve the acceptability of the tool to patients with cancer, we reduced the tool to 13 items with demonstrated validity and reliability.
  units on a scale (0-5) | 2.74 (0.93) | 2.81 (0.85) | 2.77 (0.90)

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Adherence-patient
Description: Analgesic adherence is derived from data regarding analgesics documented as prescribed (available to the patient as indicated from the medication list in the home) and analgesics consumed (from PAINReportIt). We calculate an analgesic adherence rate (dose reported as consumed divided by dose documented as prescribed, multiplied by 100) for all World Health Organization (WHO) analgesics (adjuvants, NSAIDs and non-opioids, and ATC and PRN Step 2 and Step 3 opioids).
Time Frame: Average of daily adherence (days 1 to 7)
Population: Intent to treat analysis with multiple imputation based missing data processing.
Measure: Mean (Standard Deviation); unit: proportion (0-1), higher is better
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Number analyzed (Participants) | 154 | 80
proportion (0-1), higher is better | 0.66 (0.27) | 0.67 (0.24)
Statistical Analysis 1: Comparison: Usual Hospice Care vs PAINRelieveIt (Experimental Group); Test type: Superiority; p = .43, Mixed Models Analysis

2. Secondary Outcome: Worst Pain Intensity-patient
Description: worst pain intensity in previous 24 hours measured on 0 to 10 scale where 0 means no pain and 10 means pain as bad as it can be.
Time Frame: Average of daily worse pain intensity (days 1 to 7)
Population: Intent to treat analysis with multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale (0-10); lower is better
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Number analyzed (Participants) | 154 | 80
units on a scale (0-10); lower is better | 6.05 (2.24) | 6.63 (2.12)
Statistical Analysis 1: Comparison: Usual Hospice Care vs PAINRelieveIt (Experimental Group); Test type: Superiority; p = .02, Mixed Models Analysis — Experimental group performed worse than usual care

3. Other Pre Specified Outcome: Misconceptions About Pain and Pain Management--patient
Description: Misconceptions are measured with a computer version of the Barriers Questionnaire (BQ) with response options from 0 to 5 indicating the amount of agreement with statements about barriers to pain assessment or management. Items relate to communicating with the physician about pain, side effects of analgesics, concerns about addiction, tolerance, disease progression, and being perceived as a good patient. Validity of the BQ is supported by its ability to discriminate cancer patients who report high BQ scores and also were under-medicated for their pain level and were hesitant to report their pain to their clinicians. To improve the acceptability of the tool to patients with cancer, we reduced the tool to 13 items with demonstrated validity and reliability. In prior cancer studies, patients found it to be a simple, easily understood tool that they completed in 5 minutes or less on 13 screens using a touch-screen pentablet computer.
Time Frame: pretest at baseline (day 0) & posttest on day 7; day 7 reported
Population: Intent to treat analysis with multiple imputation based missing data processing.
Measure: Mean (Standard Deviation); unit: units on a scale (0-5); lower is better
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Number analyzed (Participants) | 154 | 80
units on a scale (0-5); lower is better | 2.72 (0.79) | 2.56 (0.87)
Statistical Analysis 1: Comparison: Usual Hospice Care vs PAINRelieveIt (Experimental Group); Test type: Superiority; p = .32, Regression, Linear

4. Other Pre Specified Outcome: Satisfaction With Pain Levels -- Patient
Description: Satisfaction with pain levels is measured by two single item questions that ask the patient if he or she is satisfied with the level of pain. A three-option response allows the patient to indicate yes, no, or not sure. We tested this item in our previous study and found that 49% of patients were satisfied with their pain level at baseline were also satisfied 4 weeks later, 21% became satisfied, 18% became less satisfied and 12% were never satisfied during the 4-week study. These data are consistent with the high percentage (98%) of patients who reported a desire for no pain but whose worst pain was greater than the level they desired. Focusing on satisfaction with level of pain allows us to have greater variability in this variable than has been typically noted by other investigators.
Time Frame: Average of distribution of satisfaction with pain level reported each day (days 1 to 7).
Population: Intent to treat analysis with multiple imputation based missing data processing
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Number analyzed (Participants) | 154 | 80
Participants
  Satisfied | 50 | 24
  Not sure | 24 | 13
  Not satisfied | 80 | 43
Statistical Analysis 1: Comparison: Usual Hospice Care vs PAINRelieveIt (Experimental Group); Test type: Superiority; p = .36, Regression, Logistic

5. Other Pre Specified Outcome: Misconceptions About Pain and Pain Management--caregiver
Description: as for outcome 3
Time Frame: pretest at baseline (day 0) & posttest on day 7; day 7 reported
Population: Intent to treat analysis with multiple imputation based missing data processing.
Measure: Mean (Standard Deviation); unit: units on a scale (0-5); lower is better
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Number analyzed (Participants) | 154 | 80
units on a scale (0-5); lower is better | 2.97 (0.81) | 2.67 (0.82)
Statistical Analysis 1: Comparison: Usual Hospice Care vs PAINRelieveIt (Experimental Group); Test type: Superiority; p = .01, Regression, Linear

6. Other Pre Specified Outcome: Appropriateness of Analgesics Prescribed --Hospice Nurse
Description: We will measure the appropriateness of a patient's analgesic prescription on a given day using Cleeland's Pain Management Index (PMI). For a given day, a patient's analgesic score (0=no analgesic, 1=non-opioid, 2=weak opioid, 3=strong opioid) is subtracted by their pain intensity category (0 = worst pain of 0; 1 = worst pain of 1-3; 2 = worst pain of 4-6; 3 = worst pain of 7-10) to obtain their PMI score for the day. Negative PMI scores indicate inadequate analgesics while 0 or positive PMI scores indicate appropriate analgesics. For each patient, the outcome measure is the proportion of day with appropriate analgesics.
Time Frame: proportion of days (days 1 to 7) with appropriate analgesics
Measure: Mean (Standard Deviation); unit: proportion of days (0-1), higher=better
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
Number analyzed (Participants) | 154 | 80
proportion of days (0-1), higher=better | 0.98 (0.13) | 0.91 (0.29)
Statistical Analysis 1: Comparison: Usual Hospice Care vs PAINRelieveIt (Experimental Group); Test type: Superiority; p < 0.01, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Each patient was followed for 1 week.
Arm/Group | Usual Hospice Care | PAINRelieveIt (Experimental Group)
All-Cause Mortality (participants affected / at risk) | 14/170 | 9/92
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/92
Other Adverse Events (participants affected / at risk) | 0/170 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No